CLINICAL TRIAL: NCT00789100
Title: Evaluation of a Home-based Telemonitor Service
Brief Title: Evaluation of Remote Patient Monitoring.
Status: Withdrawn | Type: Observational
Why Stopped: Nottingham PCT withdrew for financial reasons
Sponsor: Brunel University (Other)
Collaborators: Nottingham City Primary Care Trust (Unknown)
Responsible Party: Principal Investigator, Malcolm Clarke, Reader, Brunel University
Other Study IDs: Nottingham-001
Record Dates: First submitted 2008-11-10; First posted 2008-11-11 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-07

CONDITIONS: Congestive Heart Failure; Chronic Obstructive Pulmonary Disease
Keywords: telehealth; telemonitor; telemedicine; Co-morbidities
MeSH Terms: conditions — Heart Failure; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Group provided with home-based monitor
- 2: Group receives no home-based monitor

SUMMARY:
Nottingham Primary Care Trust has launched telemonitoring to support: independent living and self-management ability of people with congestive heart failure (CHF), chronic obstructive pulmonary disease (COPD) and co-morbidities; and reduce the health care utilisation associated with these patients, including the number of hospitalisations, GP visits and community matron and specialist community nurse home visits.

The Multidisciplinary Assessment of Technology Centre for Healthcare (MATCH) will evaluate the technology and its impact of this telemonitoring system on quality of care (i.e. process measures), patient outcomes and direct healthcare costs from an NHS perspective.

DETAILED DESCRIPTION:
The study is designed to evaluate the impact of home-based monitoring to support community based nursing services and care matrons in the management of patients with CHF and COPD and co-morbidities. The main issue is to design a study that will determine the impact of the use of the technology independent of other factors. A randomised controlled trial has been chosen in which equal numbers of participants with and without home-based monitoring will be followed over the study to determine differences in utilisation of healthcare services including number of hospitalisations, length of stay in hospital, GP visits and community matron and specialist community nurse home visits.

The ethical issue is how to determine those that will receive home-based monitoring and those that will be denied. The study requires that participants are matched for severity of their condition in each arm and this could deny some from the potential benefits of monitoring. However, as only a limited number of home-based monitors are available and all participants will continue to receive normal health care services, we believe that those denied monitoring will not receive care that is different to patients not in the study and the ethical issues are acceptable.

ELIGIBILITY:
Inclusion Criteria:

* Participants selected will be those: diagnosed with CHF, COPD or co-morbidities and referred to the community management service by its selection procedure for severity of the condition; are considered eligible for home-based telemonitoring; consent to receiving telemonitoring; have an active phone connection; are able to read and speak English (language of the equipment); are capable and willing to use the home monitoring device.

Exclusion Criteria:

* Patients are considered ineligible: if they have psychological or psychiatric disorders; if they have a cognitive deficiency that makes them unable to participate in their self-treatment; if they have a visual or motor deficiency that renders them incapable of using the telemonitoring device (unless a spouse or an informal caregiver is able to help); if they are currently scheduled for a hospital admission; if their life expectancy is shorter than 2 years; or if they already participate in another study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with congestive heart failure (CHF), chronic obstructive pulmonary disease (COPD) and co-morbidities referred to the community specialist nurse or care matron
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-02; Primary Completion 2010-08 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Hospitalizations, hospital days, encounters with health professionals | Collected until end date

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Clarke, PhD, Principal Investigator — Brunel University
Locations (1):
- Nottingham PCT, Nottingham, Nottinghamshire, United Kingdom